CLINICAL TRIAL: NCT02755480
Title: Ultralow Dose Thoracic Computed Tomography in Immunocompromised Patients
Acronym: ULDCT-IC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left UHN. This study is no longer running at UHN.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-7420
Record Dates: First submitted 2015-03-12; First posted 2016-04-29 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: bone marrow transplant; infection; computed tomography; radiation dose
MeSH Terms: conditions — Leukemia; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultralow dose research (Experimental): An Ultralow Dose Thoracic Computed Tomography scan will be added to the standard of care Low dose CT scan.
  The image quality of the ultralow dose CT will be compared to the Low dose thoracic Computed Tomography.
  Interventions: Device: Ultralow Dose Thoracic Computed Tomography

INTERVENTIONS:
Device: Ultralow Dose Thoracic Computed Tomography — Ultralow dose chest CT (uLDCTT) at a radiation dose comparable to 2 chest X-rays
  Other Names: Ultralow dose CT

SUMMARY:
Patients with bone marrow cancer are more susceptible to chest infections than healthy adults; marrow ablation treatment further compromises their immune status and increases the risk of fungal opportunistic infection, which is associated with a high fatality rate. Therefore, it is critical to achieve early and accurate diagnosis of fungal infection when these patients become febrile. At the Mount Sinai Hospital (MSH) and the University Health Network (UHN), the standard of care (SOC) to exclude a chest infection in immunocompromised (IC) patients is chest computed tomography (CT) using low dose CT (LDCTT).

DETAILED DESCRIPTION:
As patients may have several febrile episodes during their hospital stay, the cumulative dose from LDCTT scans can be significant and increase the lifetime risk of inducing a second cancer. The aim of this project is to determine whether a 75% reduction in radiation dose for LDCTT in other words, an ultralow dose chest CT (uLDCTT) at a dose comparable to chest X-ray, maintains the diagnostic image quality for detection of fungal chest infection in IC patients. If successful, uLDCTT will be adopted as SOC imaging at Princess Margaret Cancer Center (PM) for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. All immunocompromised patients clinically referred for LDCTT to the Medical Imaging department at PM
2. 18 years and older

Exclusion Criteria:

1. Patients that cannot follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Image acquisition | Study Day 1
  Perform paired clinical low dose (LDCTT) and research ultralow dose (uLDCTT) chest CT in immunocompromised (IC) patients who present with febrile neutropenia (FN) and are clinically referred for LDCTT to exclude opportunistic fungal infection.

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Department of Medical Imaging, Toronto, Ontario, Canada